CLINICAL TRIAL: NCT01387620
Title: Intraindividual Randomized Clinical Comparison of DisCoVisc and Hydroxypropylmethylcellulose 2% in Phacoemulsification
Brief Title: Comparison of DisCoVisc and Hydroxypropylmethylcellulose 2%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Rodrigo França de Espíndola, MD, University of Sao Paulo - Fellow
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USP - 0111 - 09
Record Dates: First submitted 2011-06-28; First posted 2011-07-04 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2010-12

CONDITIONS: Corneal Edema; Intraocular Pressure
Keywords: Phacoemulsification; Corneal Edema; Corneal Endothelium; Viscoelastic Substances
MeSH Terms: conditions — Corneal Edema | interventions — Hyaluronic Acid; Hypromellose Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hyaluronic Acid and hydroxypropylmethylcellulose — Hyaluronic Acid 1.6% was used to performed phacoemulsification in one eye and hydroxypropylmethylcellulose 2% was used in the fellow eye.

SUMMARY:
This prospective study was performed to compare two ophthalmic viscosurgical devices, DisCoVisc (hyaluronic acid 1.6% - chondroitin sulfate 4.0%) and hydroxypropylmethylcellulose 2% in terms of their overall clinical performance during phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract
* Grade 1-3 lens opacities classification system (LOCS III)
* Pupil dilatation greater than 7.0 mm

Exclusion Criteria:

* Black, brunescent, traumatic or subluxated cataract
* Corneal endothelial disease (endothelial cell count less than 2.000 cells/mm3)
* Glaucoma, uveitis
* Previous ocular surgery

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Corneal endothelial cell count | 6 months

SECONDARY OUTCOMES:
Central Corneal Thickness | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Espindola RF, Castro EF, Santhiago MR, Kara-Junior N. A clinical comparison between DisCoVisc and 2% hydroxypropylmethylcellulose in phacoemulsification: a fellow eye study. Clinics (Sao Paulo). 2012 Sep;67(9):1059-62. doi: 10.6061/clinics/2012(09)13. PMID 23018304